CLINICAL TRIAL: NCT01269502
Title: Prevention of Secondary Foot Ulcers in Patients With Diabetes. Will People With Diabetes Who Have Had a Foot Ulcer be Able to Prevent Secondary Ulcers by Systematically Measuring Their Skin Temperature?
Brief Title: Prevention of Secondary Foot Ulcers in Patients With Diabetes Using Systematic Measuring of Skin Temperature.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 6.2009.60; 20 (Other Grant/Funding Number: Sophies Minde Ortopedi AS)
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Foot Ulcer, Diabetic
MeSH Terms: conditions — Diabetic Foot | interventions — Watchful Waiting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Skin temperature measurement (Experimental): Regular measurement of skin temperature on feet for one year
  Interventions: Device: "Temp Touch" Diabetica Solutions inc.
- Active control (Active Comparator): Daily inspection of feet for one year
  Interventions: Other: Inspection

INTERVENTIONS:
Device: "Temp Touch" Diabetica Solutions inc. — Daily measurement of skin temperature on feet for one year
  Arms: Skin temperature measurement
Other: Inspection — Inspection of feet daily for one year
  Arms: Active control

SUMMARY:
A randomised controlled pilot study on the feasibility of introducing a skin temperature device (Temp Touch) in secondary prevention of foot ulcers in people with diabetes who have had a foot ulcer in Norway.

DETAILED DESCRIPTION:
Diabetes mellitus is linked to late complications from kidneys, eyes, nerves, feet, and an increased risk of cardiovascular disease.

Approximately 170 000 people in Norway suffer from diabetes, and diabetic foot disease is one of the most common complications.

It is estimated that between 400 and 500 amputations are performed yearly in Norway, and most of the amputations are due to non-healing diabetic foot ulcers.

Efficient prevention in high-risk individuals includes follow-up in specialist foot clinics including training in self-care, adaptation of preventive footwear and insoles.

A randomised trial testing the use of skin temperature measurement in addition to routine foot care for preventing new foot ulcers showing a highly significant reduction in recurrent foot ulcers in the temperature measuring group, has previously been performed in USA (Lavery et al. Diabetes Care 2007;30:14).

This study is planned as an open, randomised pilot study of minimum 40 patients testing the feasibility of implementing the use of skin temperature measurement for prevention of recurrent diabetic foot ulcers in a specialist clinical setting in Norway.

If this is the case, we are planning a larger study to examine if these measurements can contribute to reducing the number of recurrent ulcers in clinical practice in Norway.

We are in addition using a cognitive motivational method to examine if this model can increase the use of the temperature measuring device.

ELIGIBILITY:
Inclusion Criteria:

* Previous neuropathic diabetic foot ulcer

Exclusion Criteria:

* Ankle/brachial index < 0.7. Osteomyelitis, active Charcot

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Recurrency of diabetic foot ulcer | One year

CONTACTS AND LOCATIONS:
Overall Officials: Bente K Kilhovd, Md, PhD, Principal Investigator — Oslo University Hospital Ulleval, Oslo, Norway; Anita Skafjeld, Study Chair — Oslo University Hospital, Ulleval, Oslo, Norway
Locations (1):
- Oslo university Hospital Ulleval, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Skafjeld A, Iversen MM, Holme I, Ribu L, Hvaal K, Kilhovd BK. A pilot study testing the feasibility of skin temperature monitoring to reduce recurrent foot ulcers in patients with diabetes--a randomized controlled trial. BMC Endocr Disord. 2015 Oct 9;15:55. doi: 10.1186/s12902-015-0054-x. PMID 26452544